CLINICAL TRIAL: NCT02164851
Title: Non-Invasive Shock: Differentiating Shock in the Emergency Department
Acronym: NIS
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Nathan Shapiro, Instructor of Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2013P000004
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Shock; Infection; Inflammation
Keywords: shock, emergencies, inflammation, infection; pathologic process
MeSH Terms: conditions — Shock; Infections; Inflammation; Emergencies; Pathologic Processes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 50 mLs of whole blood will be collected at enrollment for biomarker analysis
Oversight: Data Monitoring Committee: No

SUMMARY:
The goal of this study is to compare the characteristics of echocardiography and different monitoring devices in shock patients, the relationship of device parameters to biomarkers associated with shock, and determine if these any of these add clinical utility when predicting the cause of shock. We will perform a prospective, observational study of patients found to have shock physiology in the ED and follow them to determine the final shock category and ultimate outcomes.

DETAILED DESCRIPTION:
Shock is a common final pathway for many disease states, occurring when oxygen and nutrient delivery are not sufficient to maintain normal cellular function. The incidence of shock in the emergency department (ED) is approximated to be 1-3% of ED patients(1), and it carries a high mortality, ranging from 20-50% depending on the underlying cause of shock(2). Early recognition and treatment of shock significantly improves outcomes in critically ill patients(2, 3), and so the majority of efforts to this point have focused on identifying patients with shock.

The many etiologies of shock may be grouped into several broader categories: cardiogenic, distributive, hemorrhagic, hypovolemic, anaphylactic, and neurogenic. These categories cause shock through different mechanisms, but they have a significant amount of clinical overlap (4-7), making differentiating the cause of shock challenging for the emergency provider. While some overlap also exists between the treatments for these categories, several have vastly different therapeutic approaches. Since the early treatment of shock influences outcomes(2, 3, 8, 9), identifying the correct etiology to treat should logically impact outcomes as well, although this has not been studied in shock patients. However, Moore, et al., did show that physicians were only able to correctly identify the cause of hypotension in 25% of hypotensive patients in the ED, speaking to both the difficulty in diagnosing shock etiologies and the high percentage of patients with undifferentiated shock(10).

Recently, a number of different devices and biomarkers have been suggested to have clinical utility in differentiating shock and guiding resuscitation(11-13). These devices have potential to aid in the differentiation of shock.

We will conduct a prospective, observational study of patients found to have shock and "near-shock" physiology in the emergency department. We will identify patients meeting our inclusion criteria which will identify shock and "near shock" patients. Inclusion criteria will include: HR > 120, SBP < 90, or a shock index (HR/SBP) > 1 for at least five minutes. Patients that do meet vital sign requirements, but have a lactate > 4 mmol/L, will also be included.

Enrolled patients will undergo physiologic assessments using echocardiography, Microscan, Non-invasive cardiac output monitor (NICOM), and extremity temperature device, as well as a blood draw for biomarker assessment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* determined to have shock physiology, which will be defined by vital sign requirements including SBP < 90 despite appropriate resuscitation (e.g 2 L of normal saline) for at least five minutes.
* Patients that do meet vital sign requirements and vasopressor initiation will also be included

Exclusion Criteria:

* patients determined to have atrial fibrillation with rapid ventricular response or supraventricular tachycardia, and the patient is discharged when the ventricular rate is corrected.
* Patients will also be excluded if found to have to alcohol withdrawal, intoxication, or psychiatric agitation without organic cause.
* Patients with SBP < 90 mm/hg who have been documented to have chronic low blood pressure and their blood pressure is at baseline

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients found to have shock and "near-shock" physiology in the emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-11-28 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Deterioration | This measure will be assessed at the time of physician review after discharge from hospital, on average 2 months after initial ED visit.
  Composite in hospital endpoint: 1) acute renal failure (Creatinine 2x baseline or new hemodialysis), non-elective intubation, vasopressor requirement, mortality.

SECONDARY OUTCOMES:
Mortality | This measure will be assessed at the time of physician review after discharge from hospital, on average 2 months after initial ED visit.
  In-hospital mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan I Shapiro, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States